CLINICAL TRIAL: NCT03359681
Title: Perioperative Metformin Treatment for Colon Cancer, a Randomized Trial
Brief Title: Metformin Treatment for Colon Cancer
Acronym: MECORA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REG-096-2017
Record Dates: First submitted 2017-10-10; First posted 2017-12-02 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2021-11

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- metformin hydrochloride (Active Comparator): metformin, encapsulated tablet, 500mg 3 times a day for 30 days.
  Interventions: Drug: Metformin Hydrochloride
- placebo oral capsule (Placebo Comparator): placebo, encapsulated tablet, 500mg 3 times a day for 30 days.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Metformin Hydrochloride — metformin 500mg three times a day 20 days before colon cancer surgery and 10 days after.
  Other Names: metformin
  Arms: metformin hydrochloride
Drug: Placebo oral capsule — placebo 500mg three times a day 20 days before colon cancer surgery and 10 days after.
  Other Names: placebo
  Arms: placebo oral capsule

SUMMARY:
This is a double-blinded placebo controlled randomized trial examining the effect of metformin in non-diabetic patients with colon cancer on cell growth, immunological and metabolic changes. Patients are randomized to receive metformin 20 days before and 10 days after surgery. Tumor samples are examined for changes in level of cell growth and the composition of tumor cells in the tumor is examined. Blood samples are assessed for immunological markers and insulin resistance is measured. Cell proliferation, migration and adhesion are also examined in vitro by adding plasma obtained from the patients to colon cancer cell lines grown in culture.

DETAILED DESCRIPTION:
Background: Colorectal cancer (CRC) is the third most common cancer worldwide and more than 5000 patients are diagnosed each year in Denmark.

Metformin is the drug of choice for treatment of type 2 diabetes. Several studies indicate that the incidence of colorectal cancer is lower among metformin treated diabetic patients than other diabetic patients and survival after CRC is improved for this group as well.

Metformin lowers plasma glucose in diabetic patients, but studies suggest that metformin also inhibits cancer cell growth.

Tumor cell proliferation and apoptosis can be estimated by determining the expression levels of specific cell cycle related proteins such as Ki67 (proliferation) and cleaved caspase-3 (apoptosis) using immunohistochemistry.

The level of cell proliferation and apoptosis is important for tumor development, but growing evidence suggests that the microenvironment of the tumor and the patient's immune response play important roles as well. The immunoscore has been introduced as a prognostic marker for CRC. The immunoscore is determined by staining whole tumor slides for CD3 and CD8 positive lymphocytes using immunohistochemistry, followed by quantitative assessment and scoring of their densities. A high density is associated with better outcome than a low density. It is possible that metformin can influence the composition of immune cells as well.

Surgery is known to induce a surgical stress response with hormonal and metabolic changes. The stress response leads to an increased insulin resistance and hyperglycemia postoperatively. The degree of insulin resistance and hyperglycemia is correlated with risk of postoperative complications, reoperation, length of stay and death.

Study design: The trial is a randomised, placebo-controlled, double-blinded trial investigating the effect of metformin (intervention group) against placebo (control group) on cell proliferation, metabolic and immunological changes in non-diabetic patients with colon cancer.

Patients are recruited at their visit to the out-patient clinic at Slagelse Hospital when surgery is planned. Patients, who agree to participate, will be randomized to receive metformin or placebo for up to 20 days before their operation and 10 days afterwards. Blood samples will be taken at time of randomization and 4 times more during the study.

The study is divided into 5 sub-studies:

Sub-study 1 - Cell growth on tumor level: The primary outcome is determination of the difference of the level of proliferation after the intervention (time of surgery) adjusted for the level seen at baseline (time of colonoscopy). This is examined by immunohistochemical staining of tumor samples obtained from the colonoscopy and after surgery for Ki67 and cleaved caspase 3.

Sub-study 2 - immunological changes: The immunoscore is measured by immunohistochemical staining of tumor samples for CD3 and CD8 positive lymphocytes. Blood samples are analyzed for immune markers.

Sub-study 3 - cell growth in vitro: Plasma obtained from the metformin- or placebo-treated patients are added to colorectal cancer cells grown in culture. Cell proliferation, migration and adhesion are determined by in vitro studies and differences between the two groups analyzed.

Sub-study 4 - insulin resistance and recovery: Insulin resistance before and after surgery is measured using the homeostatic assessment model (HOMA) from fasting levels of glucose and insulin. Capillary glucose level is measured 4 times a day postoperatively on postoperative day 1 and 2 - before the main meals and before sleeping.

Patient perceived quality of recovery is measured using the Danish version of the validated "Quality of recovery-15" questionnaire.

Sub-study 5 - microbiota: The microbiota of fecal samples will be measured before and after metformin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with adenocarcinoma of the colon planned for elective curative intended surgery at Slagelse hospital
* Age of 18 or above
* Must be able to understand and sign informed content
* Sufficient amount of representative tumor material from the biopsies taken at the initial colonoscopy must be present

Exclusion Criteria:

* Patients diagnosed with diabetes mellitus
* Patients who are receiving or have received metformin or other oral antidiabetics
* Impaired kidney function (eGFR < 60mL/min)
* Severe liver disease (defined as transaminases above X 3 normal levels)
* Participation in another pharmacological intervention trial
* Predictable poor compliance (for instance not speaking fluent Danish, mentally impaired)
* Presenting with metastatic disease
* Patients undergoing neoadjuvant chemotherapy
* Pregnancy or lactation (fertile women must have a negative serum or urine pregnancy test to participate)
* Fertile women who do not use safe contraception during the study period.
* Allergy to metformin or placebo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Expression of Ki67 on tumor samples | colonoscopy (baseline) and at time of operation (after intervention)
  The primary outcome is determination of the difference of the level of proliferation after the intervention (time of surgery) adjusted for the level seen at baseline (time of colonoscopy). This is done using immunohistochemical staining for Ki67 (a marker for proliferation) of biopsies from the tumor. The level of proliferation will be defined as the percentage of tumor nuclei showing Ki67 staining in a specific microscopic field counted at the invasive front.

SECONDARY OUTCOMES:
Expression of cleaved Caspase-3 on tumor samples | colonoscopy (baseline) and at time of operation (after intervention)
  Determination of the difference in the level of apoptosis after the intervention (time of surgery) adjusted for the level seen at colonoscopy (baseline). Measured by immunohistochemical staining of tumor samples for cleaved Caspase-3 (marker for apoptosis).
immunoscore | time of operation (after the tumor is removed)
  At time of operation biopsies from the core and from the invasive margin of the tumor will be taken. These biopsies are stained for CD3 and CD8 positive lymphocytes and the density of these are measured.
immunological changes in bloodsamples | At baseline, day of operation and postoperative day 1, 2 and 10.
  Bloodsamples are taken at time of inclusion, day of operation and postoperative day 1,2 and 10. These are analysed for immunological markers.
insulin resistance | At the day of surgery and postoperative day 1 and 2.
  Fasting levels of glucose and insulin are measured at the day of operation (before the operation) and at postoperative day 1 and 2. Insulin resistance is measured using the HOMA-score.
blood glucose level | 4 times a day on postoperative day 1 and 2
  Blood glucose (capillary glucose) level is measured 4 times a day on postoperative day 1 and 2.
Quality of recovery | At baseline, postoperative day 1, 2, 10 and 30.
  The patients' subjective feeling of recovery is measured using the Danish version of the Quality of recovery-15 questionnaire. The questionnaire includes 15 questions with the possibility of 0 to 150 points (150 being the best possible quality of recovery)
cell growth in vitro - proliferation | At baseline, postoperative day 1 and 10.
  colon cancer cell lines will be grown in vitro in the presence of plasma from the patients. Differences in proliferation between the two groups are measured.
cell growth in vitro - adhesion | At baseline, postoperative day 1 and 10.
  colon cancer cell lines will be grown in vitro in the presence of plasma from the patients. Differences in adhesion between the two groups are measured.
cell growth in vitro - invasion | At baseline, postoperative day 1 and 10.
  colon cancer cell lines will be grown in vitro in the presence of plasma from the patients. Differences in invasion between the two groups are measured.
microbiota | At baseline and the day before surgery
  The microbiota of fecal samples will be analyzed using 16s rRNA analyses

CONTACTS AND LOCATIONS:
Overall Officials: Emilie P Colov, MD, Principal Investigator — Department of Surgery, Slagelse Hospital
Locations (1):
- Department of Surgery, Slagelse Hospital, Slagelse, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colov Tauby EP, Bojesen RD, Grube C, Miedzianogora REG, Buzquurz F, Fransgaard T, Knop FK, Gogenur I. Perioperative Metformin Treatment to Reduce Postoperative Hyperglycemia After Colon Cancer Surgery: A Randomized Clinical Trial. Dis Colon Rectum. 2024 Nov 1;67(11):1403-1412. doi: 10.1097/DCR.0000000000003426. Epub 2024 Jul 31. PMID 39437217

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT03359681/Prot_SAP_000.pdf